CLINICAL TRIAL: NCT05446545
Title: Evaluation of Prognostic and Predictive Values of Bespoke Circulating Tumor DNA Assay for Recurrent and Response Monitoring in Patients With Advanced Epithelial Ovarian Cancer
Brief Title: Bespoke ctDNA Assay for Recurrence and Treatment Response Monitoring in Advanced Epithelial Ovarian Cancer
Acronym: EOC
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: BGI Tianjin (Industry)
Responsible Party: Principal Investigator, Zhong Zheng MD, Director of Gynecologic Oncology, Fudan University
Other Study IDs: 2021-39-2342
Record Dates: First submitted 2022-04-13; First posted 2022-07-06 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; personalized ctDNA assay; treatment response monitoring; recurrence monitoring; PARPi
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ND-EOC or platinum-sensitive rEOC: 1. Newly diagnosed patients with advanced EOC (ND-EOC) who are eligible for radical surgery.
  2. Patients relapsed from platinum-based therapy (rEOC) who are eligible for secondary cytoreductive surgery.
  Interventions: Other: ND-EOC or platinum-sensitive rEOC

INTERVENTIONS:
Other: ND-EOC or platinum-sensitive rEOC — platinum-based combined chemotherapy or bevacizumab will be used for adjuvant treatment, followed by maintenance therapy with poly adenosine diphosphate-ribose polymerase (PARP) inhibitor, or bevacizumab, or other anti-tumor angiogenesis drugs or immune checkpoint inhibitors

SUMMARY:
This prospective observational study is to assess the dynamics of circulating tumor DNA (ctDNA) in patients with advanced epithelial ovarian cancer (EOC) undergoing surgery, adjuvant chemotherapy, followed by poly adenosine diphosphate-ribose polymerase (PARP) inhibitors until disease progression or the end of the study. All patients will be closely monitored throughout the course of disease by a tumor-informed bespoke ctDNA assay as well as traditional methods of surveillance, such as CA125 and imaging. This study may provide preliminary evidence for ctDNA-guided treatment decisions in future clinical practice.

DETAILED DESCRIPTION:
This observational study is designed for exploring prognostic and predictive values of the tumor-informed bespoke ctDNA assay in advanced EOC. Newly diagnosed patients who are eligible for radical surgery or relapsed patients from platinum-based adjuvant chemotherapy who are eligible for secondary cytoreductive surgery will be enrolled. The patients will be treated with SOC adjuvant therapies followed by PARP inhibitor for maintenance.

To evaluate ctDNA dynamics, tumor tissue collected from surgery will be sequenced with whole-exome sequencing (WES) to design patient-specific 16-plex panel. At planned monitoring timepoints, blood samples will be drawn, and ctDNA will be sequenced with ultra-deep ctDNA high-throughput sequencing methods.

Traditional surveillance methods will be applied as comparison, including but not limited to carbohydrate antigen 125 (CA-125)/ human epididymal protein 4 (HE4)/ carcinoembryonic antigen (CEA)/ carbohydrate antigen 199 (CA199), etc., as well as standard imaging.

Survival analyses will be conducted based on ctDNA status (positive/negative) after surgery. Recurrence rate of each subgroup, positive predictive values and negative predictive values etc. will be examined. Changes in ctDNA levels (ΔctDNA) during treatment will be used to evaluate the efficacy of maintenance therapy comparing traditional biomarkers,

ELIGIBILITY:
Inclusion Criteria:

1. Female, over 18 years of age;
2. Patients with advanced epithelial ovarian cancer who are eligible for radical surgery;
3. Patients with advanced epithelial ovarian cancer relapsed from platinum-based therapies and eligible for secondary cytoreductive surgery;
4. The subjects agree to sign the informed consent and agree to use their samples and data for related scientific research;
5. Subjects agree to collect tissue samples and peripheral blood samples for whole exon sequencing and ctDNA monitoring.

Exclusion Criteria:

1. Patients who are diagnosed, tested or treated for cancer other than ovarian cancer within 2 years (except for basal skin or squamous cell cancer that has been definitively treated);
2. Patients in pregnancy;
3. Patients with a history of blood transfusion within 3 months before enrollment;
4. Newly diagnosed patients who only received laparoscopic surgery;
5. Patients received chemotherapy or other anti-tumor therapy before surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity
Study Population: Newly diagnosed advanced EOC patients who are eligible for radical surgery or relapsed EOC patients from platinum-based adjuvant chemotherapy who are eligible for secondary cytoreductive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Two years
  Determine PFS in ctDNA positive versus ctDNA negative groups.

SECONDARY OUTCOMES:
Overall Survival (OS) | Two years
  Determine OS in ctDNA positive versus ctDNA negative groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Hao Wen, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No